CLINICAL TRIAL: NCT01074190
Title: The Effect of Neuraxial Analgesia on Maternal Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Paloma Toledo, Associate Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00007275
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Pain; Breastfeeding
Keywords: Epidural Labor Analgesia; Pain; Infant; Breastfeeding
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): spinal fentanyl 15 micrograms plus bupivacaine 2.5 mg followed by a patient controlled epidural analgesia (PCEA) maintenance infusion of bupivacaine 1mg/mL
  Interventions: Drug: Group 1
- Group 2 (Experimental): spinal fentanyl 15 micrograms plus bupivacaine 2.5 mg spinal followed by a PCEA infusion of fentanyl 1 micrograms/mL plus bupivacaine 0.8 mg/mL
  Interventions: Drug: Group 2
- Group 3 (Active Comparator): spinal fentanyl 15 micrograms plus bupivacaine 2.5mg followed by a PCEA infusion of fentanyl 2 micrograms/mL plus bupivacaine 0.625 mg/mL
  Interventions: Drug: Group 3

INTERVENTIONS:
Drug: Group 1 — A basal infusion rate for the PCEA will be set at 8 mL/h with patient administered boluses of 8 mL every 10 minutes and a one hour limit of 32 mL. Breakthrough pain in all groups will be managed using anesthesiologist administered boluses of bupivacaine 1.25 mg/mL without fentanyl.
  Other Names: bupivacaine 1mg/ml
  Arms: Group 1
Drug: Group 2 — A basal infusion rate for the PCEA will be set at 8 mL/h with patient administered boluses of 8 mL every 10 minutes and a one hour limit of 32 mL. Breakthrough pain in all groups will be managed using anesthesiologist administered boluses of bupivacaine 1.25 mg/mL without fentanyl.
  Other Names: fentanyl 1mcg/ml plus bupivacaine 0.8 mg/ml
  Arms: Group 2
Drug: Group 3 — A basal infusion rate for the PCEA will be set at 8 mL/h with patient administered boluses of 8 mL every 10 minutes and a one hour limit of 32 mL. Breakthrough pain in all groups will be managed using anesthesiologist administered boluses of bupivacaine 1.25 mg/mL without fentanyl.
  Other Names: fentanyl 2mcg/ml plus bupivacaine 0.625 mg/ml
  Arms: Group 3

SUMMARY:
A previous randomized trial showed a possible negative association with labor neuraxial analgesia with high compared to low doses of fentanyl, and breastfeeding at 6 weeks postpartum. The significance of this study would be to validate or refute these findings. In addition, we hope to better evaluate the impact of cumulative dose of fentanyl on breastfeeding success in the initial postpartum period as well as at 6 weeks and 6 months post delivery. In order to better assess the quality of breastfeeding, we will utilize a validated breastfeeding assessment tool, LATCH (Latch, Audible swallowing, Type of Nipple, Comfort, and Help). This validated tool can assess maternal and infant variables, define areas of needed intervention, and determine priorities in providing patient teaching. The LATCH assessment has been shown to be a predictor of breastfeeding duration. We also plan to vary the dosage of fentanyl analgesia to determine the relationship between doses below 150 micrograms and changes in breastfeeding assessments. If a clear association between decreased breastfeeding and total fentanyl is identified, then regimens to reduce cumulative doses of fentanyl can be developed to improve the likelihood of breastfeeding success in mothers that desire to breastfeed.

Prior observational studies have inferred epidurals negatively affect breastfeeding by decreasing maternal plasma oxytocin release which may adversely affect infant neurobehavioral development. In a study by Beilin et al., it was reported that mothers receiving a high cumulative dose (> 150 microgram) epidural fentanyl were more likely to have stopped nursing 6 weeks postpartum compared with groups receiving no fentanyl or those receiving < 150 microgram. The study however, was underpowered to detect differences in breastfeeding prior to hospital discharge. In addition, the breastfeeding assessment tool utilized resulted in binary assessments, and therefore, a global rating of the quality of breastfeeding was not available.

DETAILED DESCRIPTION:
Participants in this study will be asked to complete a questionnaire called the Intrinsic Motivation Inventory (IMI).

Subjects will be randomized at the time they request neuraxial analgesia to one of three groups: Group 1: patient controlled epidural analgesia (PCEA) with bupivacaine 1mg/mL; Group 2: PCEA with fentanyl 1 mcg/mL plus bupivacaine 0.8 mg/mL; Group 3: PCEA with fentanyl 2 mcg/mL plus bupivacaine 0.625 mg/mL. Labor analgesia will be initiated in all groups using fentanyl 15 mcg plus bupivacaine 2.5 mg administered intrathecally. A basal infusion rate for the PCEA will be set at 8 mL/h with patient administered boluses of 8 mL every 10 minutes and a one hour limit of 32 mL. Breakthrough pain in all groups will be managed using anesthesiologist administered boluses of bupivacaine 1.25 mg/mL without fentanyl.

The patient as well as individuals who evaluate the study patient will be blinded to the group assignment. Samples of maternal venous blood ½ teaspoon (2 mls) and cord blood 2ml (1/2 teaspoon) will be collected after the delivery of the fetus. Blood concentrations of fentanyl and bupivacaine will be ascertained using high performance liquid chromatography (HPLC) analysis. Success of breastfeeding using the LATCH assessment tool will be measured by the lactation nurses within 24 hrs of delivery. At 6 weeks and at 3 months postpartum, follow-up phone calls by the anesthesia service will be made to assess for duration of breastfeeding. Also, the patient's obstetrician will be contacted to obtain the patient's Edinburgh Postnatal Depression Score to assess for postpartum depression, which may be a variable in decreasing breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* English speaking
* Term gestation (> 38 weeks)
* Parous parturients presenting for attempted vaginal delivery with a cervical dilation less than 8 cm
* They must request neuraxial labor analgesia
* Have previously successfully breastfed their child postpartum for at least 6 weeks
* Are expressing an interest in exclusively breastfeeding postpartum

Exclusion Criteria:

* Under 18 years of age
* Parturients who have received parental opioids during labor or have taken opioids prenatally
* Patients whose neuraxial analgesia failed due to abnormal spinal anatomy including scoliosis or previous spinal instrumentation
* Supplemental epidural opioids during labor
* Had an expedited labor with the delivery of the fetus less than 90 minutes from the placement of the neuraxial anesthestic
* Underwent cesarean delivery
* Received general analgesia for an unanticipated postpartum procedure
* Dropout criteria include patients who wished to be taken out of the study or were lost to follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Toledo, M.D.,MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgarder DJ, Muehl P, Fischer M, Pribbenow B. Effect of labor epidural anesthesia on breast-feeding of healthy full-term newborns delivered vaginally. J Am Board Fam Pract. 2003 Jan-Feb;16(1):7-13. doi: 10.3122/jabfm.16.1.7. PMID 12583645
- [Background] Riordan J, Gross A, Angeron J, Krumwiede B, Melin J. The effect of labor pain relief medication on neonatal suckling and breastfeeding duration. J Hum Lact. 2000 Feb;16(1):7-12. doi: 10.1177/089033440001600103. PMID 11138228
- [Background] Rahm VA, Hallgren A, Hogberg H, Hurtig I, Odlind V. Plasma oxytocin levels in women during labor with or without epidural analgesia: a prospective study. Acta Obstet Gynecol Scand. 2002 Nov;81(11):1033-9. doi: 10.1034/j.1600-0412.2002.811107.x. PMID 12421171
- [Background] Beilin Y, Bodian CA, Weiser J, Hossain S, Arnold I, Feierman DE, Martin G, Holzman I. Effect of labor epidural analgesia with and without fentanyl on infant breast-feeding: a prospective, randomized, double-blind study. Anesthesiology. 2005 Dec;103(6):1211-7. doi: 10.1097/00000542-200512000-00016. PMID 16306734
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 115 | 115 | 115
Completed | 111 | 109 | 112
Not Completed | 4 | 6 | 3
Not completed — Emergency Cesarean Delivery | 1 | 2 | 1
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Delivered in under 90 minutes | 0 | 2 | 1
Not completed — Subject withdrew consent | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 111 | 109 | 112 | 332
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 109 | 112 | 332
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: Years of age] | 33 [31 to 37] | 34 [32 to 36] | 34 [31 to 36] | 34 [31 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 109 | 112 | 332
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 109 | 112 | 332
Body Mass Index (kg/m∧ 2) [Mean (Inter-Quartile Range); unit: Kilograms/meters squared] | 28 [26 to 31] | 28 [26 to 31] | 29 [26 to 31] | 28 [26 to 31]
Number of times pregnant [Mean (Inter-Quartile Range); unit: Number of times pregnant] | 3 [2 to 3] | 3 [2 to 3] | 2 [2 to 3] | 3 [2 to 3]
Live Births [Median (Inter-Quartile Range); unit: live births] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Gestational Age (Days) [Mean (Inter-Quartile Range); unit: Days] | 277 [273 to 280] | 276 [274 to 281] | 276 [273 to 279] | 276 [273 to 281]
Duration of breastfeeding with last infant [Count of Participants; unit: Participants] — Assessment of breastfeeding history with participants prior child.
  Participants
    Less than three months | 9 | 6 | 9 | 24
    3-6 months | 20 | 31 | 30 | 81
    Greater than 6 months | 82 | 72 | 73 | 227
Reason for discontinuing breastfeeding with last child [Count of Participants; unit: Participants]
  Return to work | 35 | 30 | 36 | 101
  Perceived time to stop | 22 | 22 | 20 | 64
  Lack of time | 3 | 2 | 9 | 14
  Pregnancy | 10 | 9 | 9 | 28
  Inadequate milk production | 11 | 19 | 14 | 44
  Child eating solid foods/teething | 21 | 17 | 19 | 57
  Difficulty with breastfeeding | 9 | 10 | 5 | 24
Support for breastfeeding [Count of Participants; unit: Participants]
  Weak | 0 | 2 | 1 | 3
  Moderate | 9 | 13 | 18 | 40
  Strong | 101 | 94 | 93 | 288
  Missing Data | 1 | 0 | 0 | 1
Used an assistive device/nipple shield [Count of Participants; unit: Participants]
  Used Device | 19 | 22 | 18 | 59
  Did not use device or no response | 92 | 87 | 94 | 273
Skin-to-skin contact in the first 24 hours [Count of Participants; unit: Participants]
  Did not remember | 2 | 3 | 2 | 7
  0-25% | 35 | 33 | 43 | 111
  25-50% | 28 | 41 | 39 | 108
  50-75% | 23 | 27 | 25 | 75
  75-100% | 13 | 5 | 3 | 21
  Missing Data | 10 | 0 | 0 | 10
Time from delivery to initial breastfeeding [Count of Participants; unit: Participants]
  Did not remember | 4 | 2 | 5 | 11
  0 to 1 hour | 90 | 80 | 79 | 249
  1 to 3 hours | 9 | 19 | 16 | 44
  4 to 10 hours | 4 | 4 | 5 | 13
  Greater than 10 hours | 4 | 4 | 7 | 15
Took a breastfeeding class or received breastfeeding education [Count of Participants; unit: Participants]
  Took breastfeeding class | 62 | 52 | 62 | 176
  Did not take class or no response | 49 | 57 | 50 | 156
Breastfeeding motivational measurement scale [Median (Inter-Quartile Range); unit: Score on a scale] — The breastfeeding motivational measurement tool scores the responses on a 0- poor to 140 good breastfeeding.
  Score on a scale | 119 [111 to 127] | 117 [109 to 124] | 117 [110 to 124] | 118 [109 to 127]
Verbal rating score for analgesia satisfaction (0-100) [Mean (Full Range); unit: score on a scale] — Verbal rating score for analgesia satisfaction on a scale of 0-poor to 100 good.
  score on a scale | 91 [76 to 97] | 91 [76 to 99] | 86 [74 to 96] | 89 [74 to 99]
Infant birth weight [Mean (Full Range); unit: Kilograms] | 3.54 [3.32 to 3.77] | 3.61 [3.28 to 3.91] | 3.57 [3.31 to 3.87] | 3.56 [3.28 to 3.91]
Mode of Delivery [Count of Participants; unit: Participants]
  Vaginal Delivery | 111 | 107 | 110 | 328
  Assisted Vaginal Delivery | 0 | 1 | 2 | 3
  Cesarean Delivery | 0 | 1 | 0 | 1
Breastfeeding at lactation consultant assessment n (%) [Count of Participants; unit: Participants]
  Yes | 98 | 96 | 98 | 292
  No | 8 | 9 | 3 | 20
  Consultant not available | 5 | 4 | 11 | 20
LATCH score (0-2 for each factor) [Mean (Full Range); unit: Score on scale] — LATCH is a breastfeeding charting system which provides a method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. (0- poor and 2 is good) for each section for a possible total score of 0 which is poor to 10 good.
  Score on scale
    Latch | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Audible swallowing | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Type of nipple | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Comfort (breast/nipple) | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
    Hold (positioning) | 1 [0 to 2] | 1 [1 to 1] | 1 [1 to 1] | 1 [0 to 2]
    Total Score maximum 0-10 | 8.5 [7 to 10] | 8 [6 to 10] | 9 [8 to 10] | 8.5 [6 to 10]
Skin-to-skin contact in the first 24 hours post delivery [Count of Participants; unit: Participants]
  0-25% | 72 | 70 | 71 | 213
  25-50% | 19 | 2 | 17 | 38
  50-75% | 9 | 8 | 11 | 28
  75-100% | 5 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding at 6 Weeks Post Delivery
Description: Breastfeeding continuing at 6 weeks after delivery of the baby.
Time Frame: 6 weeks post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 111 | 109 | 112
Participants
  Currently breast feeding | 100 | 99 | 102
  Not breastfeeding | 3 | 2 | 6
  Lost to follow up | 8 | 8 | 4
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority; p = .34, Chi-squared

2. Secondary Outcome: Breastfeeding at 3 Months After Delivery
Description: Breastfeeding at 3 months after delivery of baby
Time Frame: 3 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 111 | 109 | 112
Participants
  Breastfeeding | 94 | 96 | 93
  Not breastfeeding | 6 | 4 | 12
  Lost to follow up | 11 | 9 | 7
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Superiority; p = .1, Chi-squared

3. Other Pre Specified Outcome: Cumulative Fentanyl Dose (Micrograms)
Description: Total cumulative dose of fentanyl in micrograms
Time Frame: Time of epidural catheter removal
Measure: Median (Inter-Quartile Range); unit: fentalyl dose micrograms
Groups:
- Total: Cumulative Fentanyl Group 1-3
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 111 | 109 | 112 | 332
fentalyl dose micrograms | 15 [15 to 15] | 78 [60 to 109] | 139 [97 to 210] | 78 [15 to 210]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3 vs Total; A sample size of 315 achieves 80% power to detect a difference among groups using a 2 degrees of freedom Chi-Square Test with a significance level (alpha) of 0.05; Test type: Superiority; p = .1, Chi-squared

4. Other Pre Specified Outcome: Plasma Fentanyl Concentration (ng/mL)
Description: Blood plasma fentanyl concentraton (nanograms/milliliter).
Time Frame: Time of epidural catheter removal
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Total: Plasma fentanyl concentrations (ng/mL) Group 1-3
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 111 | 109 | 112 | 332
ng/mL | .01 [.007 to .02] | .07 [.05 to .09] | .13 [.09 to .18] | .07 [.007 to .18]

5. Other Pre Specified Outcome: Umbilical Vein Plasma Fentanyl Concentration (ng/mL)
Description: Umbilical venous blood plasma was analyzed for fentanyl concentration (ng/mL)
Time Frame: Immediately after delivery
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Total: Umbilical vein plasma fentanyl concentrations (ng/mL) Group 1-3
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 111 | 109 | 112 | 332
ng/mL | .005 [.005 to .1] | .03 [.02 to .04] | .06 [.04 to .09] | .03 [.005 to .09]

ADVERSE EVENTS:
Time Frame: 6 Weeks after delivery
Description: Subject contacted at 6 weeks to assess for adverse events.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/109 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/109 | 0/112
Other Adverse Events (participants affected / at risk) | 0/111 | 0/109 | 0/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=111) | Group 2 (N=109) | Group 3 (N=112)
Spinal headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) — Spinal headache reported by the subject to the study team.

LIMITATIONS AND CAVEATS:
The study was limited because few of the participants required more than 150 micrograms of fentanyl for labor analgesia. This was the cut off for reduction of breastfeeding stated by earlier studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No